CLINICAL TRIAL: NCT05398809
Title: A Phase 2 Open-Label Study to Evaluate the Efficacy and Safety of Ruxolitinib on Hair Regrowth in Patients With Autoimmune Polyendocrinopathy Candidiasis Ectodermal Dystrophy (APECED)-Associated Alopecia Areata
Brief Title: Evaluate the Efficacy and Safety of Ruxolitinib on Hair Regrowth in Patients With Autoimmune Polyendocrinopathy Candidiasis Ectodermal Dystrophy (APECED)-Associated Alopecia Areata
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000861; 000861-I
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11-26

CONDITIONS: Autoimmune Polyendocrinopathy Candidiasis Ectodermal Dystrophy (Apeced); Alopecia Areata
Keywords: Aps-1; Aire; Jak; Autiommunity; Hair Loss
MeSH Terms: conditions — Polyendocrinopathies, Autoimmune; Alopecia Areata; Alopecia | interventions — ruxolitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib/APECED-AA Patients (Experimental): All participants receiving IP through this protocol (APECED-AA patients)will receive ruxolitinib.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib (Jakafi) is approved by the FDA for the treatment of intermediate or high-risk myelofibrosis in adults, polycythemia vera in adults who have had an inadequate response to or are intolerant of hydroxyurea, and acute and chronic graft-versus-host disease in adult and pediatric patients (aged =12 years).

SUMMARY:
Background:

Autoimmune polyendocrinopathy candidiasis ectodermal dystrophy (APECED) is a problem of the immune system. In people with APECED, the immune system makes a mistake and attacks the body. Some people with APECED have a type of hair loss called alopecia areata (AA). No drugs are approved to treat AA.

Objective:

To see if a study drug (ruxolitinib) can help hair regrowth in people with APECED-associated AA and if it can improve other symptoms caused by the immune system s attack to the body.

Eligibility:

People aged 12 to 65 years with APECED and severe AA.

Design:

Participants will be in this study for up to 10 months. They will have 5 in-person visits and 6 televisits, each about 4 weeks apart. One in-person visit may be up to a 10-day stay in the hospital.

The first in-person visit will include screening. Participants will have a physical exam. They will have blood tests. Photographs may be taken of their skin. They will answer questions about their quality of life.

Participants will begin taking the study drug during their hospital stay. They will take the pills by mouth twice a day for 8 months. Researchers may take tissue samples from participants scalp, gums, and lower lip. Participants may provide samples of urine, stool, nail clippings, and saliva. They may have an eye exam and an ultrasound exam of their abdomen.

Some tests may be repeated in subsequent in-person visits.

In telehealth visits, participants will answer questions about how they are feeling. They will describe and send photos of hair regrowth. They will be asked to have blood drawn and the results sent to the researchers.

DETAILED DESCRIPTION:
Study Description:

This is a phase 2 open-label study to evaluate the efficacy and safety of the Janus-associated kinase (JAK) inhibitor, ruxolitinib, in severe APECED-associated alopecia areata (AA). Following an 8-week observation period to assess baseline disease state, qualifying participants may be admitted for up to 10 days for an inpatient visit to start receiving twice daily dosing of oral ruxolitinib. The dose will be increased at weeks 8 and 16, but may be maintained or reduced if the participant experiences certain adverse events (AEs). The total duration of the ruxolitinib regimen is 8 months. At in-person study visits, participants will be monitored for AEs/reactions and will complete patient-reported outcome (PRO) metrics to track their symptoms and general wellbeing. Participants will also have televisits during the months when there is no in-person visit, for AE assessment and local blood draws for safety labs.

Family members or household contacts of participants will also be enrolled to complete a quality-of-life survey, for comparison with a corresponding patient survey.

Primary Objective:

To evaluate the efficacy of ruxolitinib on hair regrowth in participants with APECED-associated AA.

Secondary Objectives:

1. To evaluate the safety of ruxolitinib in patients with APECED-associated AA.
2. To assess additional measures of efficacy related to hair regrowth in response to ruxolitinib treatment.
3. To investigate the effect of ruxolitinib on PROs related to hair regrowth.
4. To evaluate the effect of ruxolitinib on histologic and immunologic features of the skin.

Exploratory Objectives:

1. To investigate the effect of ruxolitinib on improving clinical symptoms and associated laboratory, histologic, and immunologic abnormalities in affected organs and tissues beyond the skin.
2. To investigate the effect of ruxolitinib on PROs of affected organs and tissues beyond the skin.
3. To investigate the effect of ruxolitinib on prevention of development of new APECED associated complications during the 32-week treatment period.
4. To examine the effects of ruxolitinib on ameliorating immunologic readouts of excessive interferon (IFN)- >=/JAK/STAT signaling in peripheral blood and affected organs and tissues beyond the skin.
5. To determine whether ruxolitinib treatment affects the composition of microbial communities at the mucocutaneous barriers.

Primary Endpoint:

Response defined as a 30 percent improvement from baseline in the Severity of Alopecia Tool (SALT) score at 32 weeks.

Secondary Endpoints:

1. Incidence of SAEs, AEs requiring study drug discontinuation, and other AEs.
2. Achievement of 30 percent improvement of SALT score (SALT30) at week 16.
3. Achievement of 50 percent improvement of SALT score (SALT50) at week 32.
4. Achievement of SALT score <=20 at week 32.
5. Time for participants to achieve SALT score <=20.
6. Time for participants to achieve SALT30 and SALT50.
7. Percentage of hair regrowth at week 32.
8. Improvement of Alopecia Areata Symptom Impact Scale (AASIS) score from baseline at week 32.
9. Improvement of Dermatology Life Quality Index (DLQI) score (adults) from baseline at week 32.
10. Improvement of Children s Dermatology Life Quality Index (CDLQI) score (pediatrics) from baseline at week 32.
11. Improvement of Family Dermatology Life Quality Index (FDLQI) score (family members or household contacts) from baseline at week 32.
12. Improvement of the 36-Item Short Form Survey (SF-36) score (adults) from baseline at week 32.
13. Improvement of the Pediatric Quality of Life Inventory (PedsQL) score (pediatrics) from baseline at week 32.
14. PRO for Scalp Hair Assessment Score of 0 or 1 with a >=2-point improvement from baseline among participants with a score of >=3 at baseline at week 32.
15. Improvement of AA investigator global assessment (IGA) measure from baseline at week 32.
16. Achievement of clinician-reported outcome (ClinRO) measure for eyebrow (EB) hair loss 0 or 1 with >=2-point improvement from baseline (among participants with ClinRO measure for EB hair loss >=2 at baseline) at week 32.
17. Achievement of ClinRO measure for eyelash (EL) hair loss 0 or 1 with >=2-point improvement from baseline (among participants with ClinRO measure for EL hair loss 2 at baseline) at week 32.
18. Change from baseline in Skindex-16 AA symptoms, emotions, and functioning domain scores at week 32.
19. Change from baseline in histologic and immunologic abnormalities of scalp tissue at week 32.

Exploratory Endpoints:

1. Change from baseline in histologic or immunologic abnormalities of salivary gland tissue in participants with Sj(SqrRoot)(Delta)gren s-like syndrome at week 32.
2. Change from baseline in histologic or immunologic abnormalities of oral mucosal tissue at week 32.
3. Change from baseline in histologic or immunologic abnormalities of gastric tissue in participants with gastritis at week 32.
4. Change from baseline in histologic or immunologic abnormalities of duodenal tissue in participants with intestinal dysfunction at week 32.
5. Time to development of next APECED-associated manifestation(s) over the 32-week treatment period.
6. Number of APECED-associated manifestations developed over the 32-week treatment period.
7. Development of new APECED-associated manifestation(s) over the 32-week treatment period.
8. Change from baseline in irritable bowel syndrome (IBS) quality of life (QOL) and small intestinal bacterial overgrowth (SIBO) questionnaire scores in participants with intestinal dysfunction at week 32.
9. Change from baseline in salivary flow rate in participants with Sj(SqrRoot)(Delta)gren s-like syndrome at week 32.
10. Change from baseline in corticosteroid dose requirements, adrenocorticotropic hormone, cortisol, electrolyte, and renin levels in participants with adrenal insufficiency at week 32.
11. Change from baseline in thyroid hormone replacement dose requirements, thyroid-stimulating hormone (TSH), free and total thyroxine, anti-thyroglobulin, and thyroid peroxidase antibody in participants with hypothyroidism at week 32.
12. Change from baseline in calcium replacement requirements, intact parathyroid hormone, and calcium levels in participants with hypoparathyroidism.
13. Change from baseline in insulin requirements, hemoglobin A1C (HbA1c), fasting glucose, insulin, c-peptide, urine ketone, and glucose levels in participants with type 1 diabetes at week 32.
14. Change from baseline in levels of follicle-stimulating hormone, estradiol, Anti-Mullerian hormone, total and free testosterone, and sex hormone binding globulin in participants with hypogonadism at week 32.
15. Change from baseline in vitamin B12 and intrinsic factor antibody levels in participants with pernicious anemia at week 32.
16. Change from baseline in Vitiligo Area Scoring Index (VASI) in participants with vitiligo at week 32.
17. Change from baseline in Ocular Surface Disease Index score (OSDI) in participants with dry eyes at week 32.
18. Change from baseline measure corneal fluorescein staining (grading scale), tear breakup time (TBUT, in seconds), automated keratography TBUT, and tear meniscus assessments in participants with keratoconjunctivitis at week 32.
19. Change from baseline grade of conjunctival redness in participants with keratoconjunctivitis at week 32.
20. Change from baseline in tear production as assessed by Schirmer s test in participants with Sj(SqrRoot)(Delta)gren s-like syndrome at week 32.
21. Change from baseline in frequency and severity for oral, vaginal, and/or nail candidiasis during the 32-week treatment period.
22. Change from baseline in spleen volume as measured by ultrasound at week 32.
23. Change from baseline in nail appearance in participants with nail dystrophy at week 32.
24. Improvement in ClinRO PRO for nail appearance from baseline at 32 weeks.
25. Change from baseline in cytokine- and tissue-specific autoantibodies over the 32-week treatment period.
26. Change from baseline of levels of phosphorylated STAT molecules in peripheral blood mononuclear cells (PBMCs) over the 32-week treatment period.
27. Change from baseline in serum levels of IFN-Y, CXCL9, CXCL10, and/or other immune-based biomarkers over the 32-week treatment period.
28. Change from baseline in transcriptional profile in whole blood and tissue biopsies over the 32-week treatment period.
29. Change from baseline in the oral, vaginal, stool, and/or skin microbiome over the 32-week treatment period.

ELIGIBILITY:
* INCLUSION CRITERIA:

For participants with APECED-associated AA:

1. Participant must be able to understand and provide informed consent.
2. Aged >=12 to <=75 years.
3. Patients with APECED (genetic or clinical diagnosis) and severe AA (defined as having >=50% total scalp loss at screening per the SALT score).
4. Duration of hair loss greater than 6 months.
5. No present evidence of hair regrowth.
6. Is na(SqrRoot) ve or unresponsive to other treatments for AA.
7. No treatment for alopecia in the past 2 months prior to study enrollment.
8. Willingness to use valacyclovir prophylaxis for the prevention of herpes viral reactivation.
9. Vaccinations should be up to date in agreement with current CDC immunization guidelines prior to start of ruxolitinib.
10. Proficient in written English.
11. Participants who can get pregnant or impregnate their partner must agree to use at least one highly effective method of contraception when engaging in sexual activities that can result in pregnancy, starting at screening until 12 weeks after the last dose. Highly effective contraceptive measures include:

    1. Stable use of combined (estrogen- and progestogen-containing) hormonal contraception (oral, intravaginal, transdermal) or progestogen-only hormonal contraception (oral, injectable, implantable) starting 1 month prior to screening.
    2. Intrauterine device; intrauterine hormone-releasing system.
    3. Two barrier methods (eg, condom with spermicide, diaphragm with spermicide, or cervical cap and spermicide). Internal and external condoms may not be used together.
    4. Bilateral tubal ligation.

Periodic abstinence (calendar, symptothermal, and post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method are not acceptable methods of contraception.

For family members or household contacts:

1. Aged >=18 years.
2. Lives with the participant.
3. Proficient in written English.

EXCLUSION CRITERIA:

For participants with APECED-associated AA:

1. Known history of hypersensitivity to ruxolitinib or other JAK inhibitors.
2. History of or active skin disease on the scalp other than AA, such as psoriasis or seborrheic dermatitis.
3. Diagnosis of AA is in question or the pattern of hair loss is such that quantification of hair loss and assessment of regrowth is difficult, eg, patients with androgenic alopecia.
4. Treated within the last 2 months with intralesional steroids, systemic steroids, anthralin, squaric acid, diphenylcyclopropenone, tacrolimus, minoxidil, or other medication that, in the opinion of the investigator, may affect hair regrowth.
5. Current or recent use of any investigational drug (within 3 months or 5 half-lives, whichever is longer, prior to screening).
6. Scheduled to participate in another clinical study involving an investigational drug during the course of this study.
7. Use of systemic immunosuppressive or immune-modulating agents within 3 months prior to screening, except systemic steroids 10 mg of prednisone equivalent per day.
8. Current use of systemic steroids with daily dose >10 mg of prednisone equivalent for any reason or steroid burst for >3 days within 1 month of screening.
9. History of alcohol or drug abuse within 6 months prior to screening.
10. Presence of one or more of the following clinically significant laboratory abnormalities:

    1. Serum ALT>=3 times upper limit of normal (ULN).
    2. Serum total bilirubin >=2 times ULN.
    3. ANC<=1000 cells/microliter.
    4. Hemoglobin <=9.0 g/dL.
    5. Platelet count <=100,000/microliter.
    6. Serum creatinine >=2 times ULN.
11. Planned or anticipated major surgical procedure during the study.
12. Plans to receive any live vaccines within 1 month of the anticipated first dose of ruxolitinib.
13. Known or suspected immunodeficiency disorder besides APECED.
14. History of untreated invasive opportunistic infections (eg, tuberculosis, non-tuberculous mycobacterial infections, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystis pneumonia, aspergillosis) despite infection resolution or otherwise recurrent infections of

    abnormal frequency or prolonged infections suggesting an immune-compromised status as judged by the investigator.
15. Untreated latent tuberculosis infection.
16. Infection with HIV.
17. Untreated infection with hepatitis B or C.
18. History of serious bacterial infection within the last 3 months prior to screening, unless treated and resolved with antibiotics, or any chronic bacterial infection (eg, chronic pyelonephritis, osteomyelitis).
19. History of unprovoked DVT, PE, arterial thrombosis, or other thrombotic events.
20. History of stroke, heart attack, or heart failure.
21. History of herpes zoster or cytomegalovirus infection that resolved within 2 months prior to screening.
22. History of basal cell carcinoma, localized squamous cell carcinoma of the skin, or in situ carcinoma of the cervix, unless the participant is in remission and curative therapy was completed at least 12 months prior to screening.
23. History of other malignancies, unless the participant is in remission and curative therapy was completed at least 5 years prior to screening.
24. Planned or anticipated use of any prohibited medications and procedures during the study.
25. Current pregnancy or breastfeeding.
26. Past or current medical problems or findings from physical examination, EKG, or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant s ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

There are no exclusion criteria for family members or household contacts.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Response defined as a 30% improvement from baseline in the Severity of Alopecia Tool (SALT) score at 32 weeks. | 32 weeks
  To evaluate the efficacy of ruxolitinib on hair regrowth in participants with APECED-associated AA

SECONDARY OUTCOMES:
Improvement of AA-IGA measure from baseline at week 32. | Week 32
  1. To evaluate the safety of ruxolitinib in patients with APECED associated AA 2. Assess additional measures of efficacy related to hair regrowth in response to ruxolitinib treatment. 3. Investigate the effect of ruxolitinib on PROs related to hair regrowth. 4. Evaluate the effect of ruxolitinib on the histologic and immunologic features of the skin.
Improvement of DLQI score (adults) from baseline at week 32. | Week 32
  1. To evaluate the safety of ruxolitinib in patients with APECED associated AA 2. Assess additional measures of efficacy related to hair regrowth in response to ruxolitinib treatment. 3. Investigate the effect of ruxolitinib on PROs related to hair regrowth. 4. Evaluate the effect of ruxolitinib on the histologic and immunologic features of the skin.
Improvement of AASIS score from baseline at week 32. | Week 32
  1. To evaluate the safety of ruxolitinib in patients with APECED associated AA 2. Assess additional measures of efficacy related to hair regrowth in response to ruxolitinib treatment. 3. Investigate the effect of ruxolitinib on PROs related to hair regrowth. 4. Evaluate the effect of ruxolitinib on the histologic and immunologic features of the skin.
Percentage of hair regrowth at week 32. | Week 32
  1. To evaluate the safety of ruxolitinib in patients with APECED associated AA 2. Assess additional measures of efficacy related to hair regrowth in response to ruxolitinib treatment. 3. Investigate the effect of ruxolitinib on PROs related to hair regrowth. 4. Evaluate the effect of ruxolitinib on the histologic and immunologic features of the skin.
Time for participants to achieve SALT30 and SALT50. | Variable
  1. To evaluate the safety of ruxolitinib in patients with APECED associated AA 2. Assess additional measures of efficacy related to hair regrowth in response to ruxolitinib treatment. 3. Investigate the effect of ruxolitinib on PROs related to hair regrowth. 4. Evaluate the effect of ruxolitinib on the histologic and immunologic features of the skin.
Achievement of SALT50 at week 32. | Week 32
  1. To evaluate the safety of ruxolitinib in patients with APECED associated AA 2. Assess additional measures of efficacy related to hair regrowth in response to ruxolitinib treatment. 3. Investigate the effect of ruxolitinib on PROs related to hair regrowth. 4. Evaluate the effect of ruxolitinib on the histologic and immunologic features of the skin.
Achievement of SALT30 at week 16. | Week 16
  1. To evaluate the safety of ruxolitinib in patients with APECED associated AA 2. Assess additional measures of efficacy related to hair regrowth in response to ruxolitinib treatment. 3. Investigate the effect of ruxolitinib on PROs related to hair regrowth. 4. Evaluate the effect of ruxolitinib on the histologic and immunologic features of the skin.
Change from baseline in histologic and immunologic abnormalities of scalp tissue at week 32. | Week 32
  1. To evaluate the safety of ruxolitinib in patients with APECED associated AA 2. Assess additional measures of efficacy related to hair regrowth in response to ruxolitinib treatment. 3. Investigate the effect of ruxolitinib on PROs related to hair regrowth. 4. Evaluate the effect of ruxolitinib on the histologic and immunologic features of the skin.
Change from baseline in Skindex-16 AA symptoms, emotions, and functioning domain scores at week 32. | Week 32
  1. To evaluate the safety of ruxolitinib in patients with APECED associated AA 2. Assess additional measures of efficacy related to hair regrowth in response to ruxolitinib treatment. 3. Investigate the effect of ruxolitinib on PROs related to hair regrowth. 4. Evaluate the effect of ruxolitinib on the histologic and immunologic features of the skin.
Achievement of ClinRO measure for EL hair loss 0 or 1 with =2-point improvement from baseline (among participants with ClinRO measure for EL hair loss =2 at baseline) at week 32. | Week 32
  1. To evaluate the safety of ruxolitinib in patients with APECED associated AA 2. Assess additional measures of efficacy related to hair regrowth in response to ruxolitinib treatment. 3. Investigate the effect of ruxolitinib on PROs related to hair regrowth. 4. Evaluate the effect of ruxolitinib on the histologic and immunologic features of the skin.
16. Achievement of ClinRO measure for EB hair loss 0 or 1 with =2-point improvement from baseline (among participants with ClinRO measure for EB hair loss =2 at baseline) at week 32. | Week 32
  1. To evaluate the safety of ruxolitinib in patients with APECED associated AA 2. Assess additional measures of efficacy related to hair regrowth in response to ruxolitinib treatment. 3. Investigate the effect of ruxolitinib on PROs related to hair regrowth. 4. Evaluate the effect of ruxolitinib on the histologic and immunologic features of the skin.
PRO for Scalp Hair Assessment Score of 0 or 1 with a =2-point improvement from baseline among participants with a score of =3 at baseline at week 32. | Week 32
  1. To evaluate the safety of ruxolitinib in patients with APECED associated AA 2. Assess additional measures of efficacy related to hair regrowth in response to ruxolitinib treatment. 3. Investigate the effect of ruxolitinib on PROs related to hair regrowth. 4. Evaluate the effect of ruxolitinib on the histologic and immunologic features of the skin.
Improvement of PedsQL score (pediatrics) from baseline at week 32. | Week 32
  1. To evaluate the safety of ruxolitinib in patients with APECED associated AA 2. Assess additional measures of efficacy related to hair regrowth in response to ruxolitinib treatment. 3. Investigate the effect of ruxolitinib on PROs related to hair regrowth. 4. Evaluate the effect of ruxolitinib on the histologic and immunologic features of the skin.
Improvement of SF-36 score (adults) from baseline at week 32. | Week 32
  1. To evaluate the safety of ruxolitinib in patients with APECED associated AA 2. Assess additional measures of efficacy related to hair regrowth in response to ruxolitinib treatment. 3. Investigate the effect of ruxolitinib on PROs related to hair regrowth. 4. Evaluate the effect of ruxolitinib on the histologic and immunologic features of the skin.
Improvement of FDLQI score (family members or household contacts) from baseline at week 32. | Week 32
  1. To evaluate the safety of ruxolitinib in patients with APECED associated AA 2. Assess additional measures of efficacy related to hair regrowth in response to ruxolitinib treatment. 3. Investigate the effect of ruxolitinib on PROs related to hair regrowth. 4. Evaluate the effect of ruxolitinib on the histologic and immunologic features of the skin.
Improvement of CDLQI score (pediatrics) from baseline at week 32. | Week 32
  1. To evaluate the safety of ruxolitinib in patients with APECED associated AA 2. Assess additional measures of efficacy related to hair regrowth in response to ruxolitinib treatment. 3. Investigate the effect of ruxolitinib on PROs related to hair regrowth. 4. Evaluate the effect of ruxolitinib on the histologic and immunologic features of the skin.
Incidence of SAEs, AEs requiring study drug discontinuation, and other AEs. | End of Study
  1. To evaluate the safety of ruxolitinib in patients with APECED associated AA 2. Assess additional measures of efficacy related to hair regrowth in response to ruxolitinib treatment. 3. Investigate the effect of ruxolitinib on PROs related to hair regrowth. 4. Evaluate the effect of ruxolitinib on the histologic and immunologic features of the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Michail S Lionakis, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000861-I.html